CLINICAL TRIAL: NCT06797869
Title: Efficacy and Safety of co Administered Cagrilintide and Semaglutide (CagriSema) Once Weekly Versus Placebo in Participants With Type 2 Diabetes and Painful Diabetic Peripheral Neuropathy
Brief Title: A Research Study to Investigate the Effects of CagriSema Compared to Placebo in People With Type 2 Diabetes and Painful Diabetic Peripheral Neuropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-7864; U1111-1306-9422 (Other: World Health Organization (WHO)); 2023-509662-38 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-01-27; First posted 2025-01-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Participants will receive CagriSema (Cagrilintide B + Semaglutide I) subcutaneously once weekly for 32 weeks.
  Interventions: Drug: CagriSema (Cagrilintide B and Semaglutide I)
- Placebo (Placebo Comparator): Participants will receive placebo matched to CagriSema (Cagrilintide B + Semaglutide I) subcutaneously once weekly for 32 weeks.
  Interventions: Drug: Placebo matched to CagriSema (Cagrilintide B and Semaglutide I)

INTERVENTIONS:
Drug: CagriSema (Cagrilintide B and Semaglutide I) — Cagrilintide B and Semaglutide I will be administered subcutaneously using DV3384 pen-injector.
  Arms: CagriSema
Drug: Placebo matched to CagriSema (Cagrilintide B and Semaglutide I) — Placebo matched to Cagrilintide B and Placebo matched to Semaglutide I will be administered subcutaneously using DV3384 pen-injector.
  Arms: Placebo

SUMMARY:
This study will look at the effects of CagriSema in people with both type 2 diabetes and painful diabetic peripheral neuropathy, compared to placebo. Participants will either get an active medicine or a "dummy" medicine (placebo). Which treatment participants get is decided by chance. In this study the active, investigational medicine is called CagriSema. Doctors cannot yet prescribe CagriSema. For each participant, the study will last for about 10 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female.
* Age 18 years or above at the time of signing the informed consent.
* Body mass index (BMI) ≥25.0 kilogram per square meter (kg/m^2) at screening.
* Diagnosis of type 2 diabetes (T2D) ≥180 days before screening.

  -- For participants on anti-diabetic drugs: Stable daily and/or weekly dose(s) ≥90 days before screening of any of the following anti-diabetic drug(s) or combination regimen(s) at effective or maximum tolerated dose, as judged by the investigator:
  * Treatment with 1-3 marketed oral anti-diabetic drugs (OADs) (metformin, α-glucosidase inhibitors (AGI), glinides, sodium-glucose co-transporter 2 inhibitors (SGLT2i), thiazolidinediones, or sulphonylureas (SU) as a single agent or in combination) according to local guidelines.
  * Treatment with basal or basal-bolus insulin (including premixed insulin formulations) according to local guidelines.
* HbA1c ≤10.5 % (91 millimole per mole [mmol/mol]) and ≥6.0 % (42 mmol/mol), as determined by central laboratory at screening.
* Diagnosis of painful diabetic peripheral neuropathy (pDPN) at screening as well as at the following criteria:

  -- Participant with self-reported pain consistent with pDPN for a minimum of 3 months before screening, as judged by the investigator.
* Stable pharmacological and non-pharmacological treatment of pain for a minimum of 3 months before screening, in the opinion of the investigator. The treatment regimen should adhere to local guidelines (if available).

Key Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Use of any glucagon-like peptide-1 receptor agonist (GLP-1 RA), including medication with GLP-1 RA activity, (DPP-4), or amylin analogue within 60 days before screening.
* Significant use of opioids, cannabinoids or benzodiazepines within 30 days before screening, in the opinion of the investigator. Significant use is defined as use that renders it unlikely that the participant is able to comply with protocol requirements for discouraged medications.
* Anticipated initiation or clinically relevant change in concomitant medications (for more than 14 consecutive days during the study) known to affect weight or glucose metabolism (e.g., orlistat, thyroid hormones or oral corticosteroids).
* Planned initiation or change in anti-depressant, anti-psychotic or anti-epileptic medication. If participants are already taking such medication, they should have stable and optimised treatment for at least 8 weeks before screening.
* Presence or history of epilepsy and fibromyalgia.
* Presence of non-diabetic neuropathies, in the opinion of the investigator.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination and OCT assessment performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Any other painful medical condition(s) where the pain is significantly more severe than the diabetic peripheral neuropathy pain, as judged by the investigator (participants will not be excluded if the pain is transient in nature).
* History of suicidal attempt within 5 years before screening
* Suicidal behaviour within 1 month before screening.
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) <30 ml/min/1.73 m2 as determined by central laboratory at screening.
* Exposure to an investigational medicinal product within 90 days or 5 half-lives of the investigational medicinal product (if known), whichever is longer, before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Change in weekly average Pain Intensity-Numerical Rating Scale (PI-NRS) | From baseline (week 0) to end of treatment (week 32)
  Measured as score on a scale.

SECONDARY OUTCOMES:
Number of participants reaching ≥30 percentage (%) reduction in PI-NRS | From baseline (week 0) to end of treatment (week 32)
  Measured as count of participants.
Time to achieve ≥30% reduction in weekly average PI-NRS | From baseline (week 0) to end of treatment (week 32)
  Measured as days.
Number of participants reaching ≥50 % reduction in PI-NRS | From baseline (week 0) to end of treatment (week 32)
  Measured as count of participants.
Time to achieve ≥50% reduction in weekly average PI-NRS | From baseline (week 0) to end of treatment (week 32)
  Measured as days.
Change in Brief Pain Inventory-Short Form (BPI-SF) | From baseline (week 0) to end of treatment (week 32)
  Measured as score on a scale.
Change in Chronic Pain Sleep Inventory 3-item (CPSI 3) | From baseline (week 0) to end of treatment (week 32)
  Measured as score on a scale.
Change in Michigan Neuropathy Screening Instrument (MNSI) | From baseline (week 0) to end of treatment (week 32)
  Measured as score on a scale.
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 32)
  Measured as millimeters of mercury (mmHg).
Change in diastolic blood pressure | From baseline (week 0) to end of treatment (week 32)
  Measured as mmHg.
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 32)
  Measured as percentage of HbA1c.
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 32)
  Measured as millimole per liter (mmol/L).
Relative change in body weight | From baseline (week 0) to end of treatment (week 32)
  Measured as percentage change.
Change in waist circumference | From baseline (week 0) to end of treatment (week 32)
  Measured as centimeter (cm).
Ratio to Baseline in Lipids: Total Cholesterol | From baseline (week 0) to end of treatment (week 32)
  Measured as ratio.
Ratio to Baseline in Lipids: High-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 32)
  Measured as ratio.
Ratio to Baseline in Lipids: Low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 32)
  Measured as ratio.
Ratio to Baseline in Lipids: Very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 32)
  Measured as ratio.
Ratio to Baseline in Lipids: Triglycerides | From baseline (week 0) to end of treatment (week 32)
  Measured as ratio.
Ratio to Baseline in Lipids: Free fatty acids | From baseline (week 0) to end of treatment (week 32)
  Measured as ratio.
Ratio to Baseline in Lipids: Non-HDL cholesterol | From baseline (week 0) to end of treatment (week 32)
  Measured as ratio.
Relative change in high sensitivity C-reactive protein (hsCRP) | From baseline (week 0) to end of treatment (week 32)
  Measured as percentage change.
Number of treatment-emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 38)
  Measured as count of events.
Number of treatment-emergent serious adverse events (TESAEs) | From baseline (week 0) to end of study (week 38)
  Measured as count of events.
Number of severe hypoglycaemic episodes (level 3) (No specific glucose threshold) | From baseline (week 0) to end of study (week 38)
  Severe hypoglycaemia is a severe event characterised by altered mental and/or physical status requiring assistance from another person to actively administer carbohydrates, glucagon, or take other corrective actions to treat hypoglycaemia. Measured as count of episodes.
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL) confirmed by blood glucose meter)) | From baseline (week 0) to end of study (week 38)
  Measured as count of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (54):
- United States (19):
  - eStudySite, La Mesa, California
  - Linda Vista Health Care Ctr, San Diego, California
  - My Preferred Research, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Foot & Ankle Center of Illinois, Springfield, Illinois
  - Velocity Clinical Research Rockville, Rockville, Maryland
  - Amicis Centers of Clinical Research, St Louis, Missouri
  - DM Clinical - CyFair, Albuquerque, New Mexico
  - Southgate Medical Group, LLP, West Seneca, New York
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Oregon Health & Science University, Portland, Oregon
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - DM Clinical - CyFair, Houston, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - DM Clinical - CyFair, San Antonio, Texas
  - DM Clinical Research, San Antonio, Texas
  - Velocity Clinical Research Portsmouth, Suffolk, Virginia
- Canada (7):
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Centricity Research Brampton, Brampton, Ontario
  - Centricity Clinical Research Burlington, Burlington, Ontario
  - Centricity Research Etobicoke, Etobicoke, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
- Denmark (5):
  - Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus N
  - Steno Diabetes Center Nordjylland, Gistrup
  - Steno Diabetes Center Copenhagen, Herlev
  - Kolding Sygehus Karkirurgi, Kolding
  - Steno Diabetes Center Odense, Odense C
- France (5):
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Groupe Sos Sante-Hopital Le Creusot-Hotel Dieu-1, Le Creusot
  - Aphp-Hopital La Pitie Salpetriere-1, Paris
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque-1, Pessac
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Norway (4):
  - Haukeland Universitetssykehus, Bergen
  - Sykehuset Innlandet HF Hamar, Hamar
  - Oslo universitetssykehus, Ullevål, Oslo
  - Stavanger Universitetssykehus, Helse Stavanger HF, Stavanger
- Spain (7):
  - Hospital Nisa Sevilla Aljarafe, Castilleja de La Cuesta. Sevilla, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Infanta Luisa, Seville
- United Kingdom (7):
  - Tameside General Hospital, Ashton-under-Lyne, Greater Manchester
  - Ipswich Hospital - Diabetes, Ipswich
  - Aintree University Hospital, Liverpool
  - St Pancras Clinical Research, London
  - Kings College Hospital - Renal, London
  - Manchester Royal Infirmary - Diabetes, Manchester
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com